CLINICAL TRIAL: NCT00865488
Title: A Prospective, Controlled, Randomized, Multi-Center, Pivotal Study Evaluating the Safety and Efficacy of AdhexilTM in Prevention And/Or Reduction of Adhesions in Gynecology Surgery
Brief Title: Evaluation of Adhexil Safety and Efficacy in Prevention and/or Reduction of Adhesions in Gynecological Surgery
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Eran Kurman, Clinical Affairs Manager, Omrix Biopharmaceuticals Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AA-GYN-002
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Ovarian Cysts; Endometriosis; Adhesions
MeSH Terms: conditions — Ovarian Cysts; Endometriosis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): patients who will be treated in accordance with standard of care
- 2 (Experimental): patients for which Adhexil will be applied to prevent/reduce adhesions
  Interventions: Biological: ADHEXIL

INTERVENTIONS:
Biological: ADHEXIL — Adhesions prevention
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ADHEXIL™ in preventing and/or reducing post-operative adhesions in patients undergoing surgery involving the ovaries.

DETAILED DESCRIPTION:
Patients will be divided into two arms: 1) patients who will be treated in accordance with standard of care; 2) patients for which ADHEXIL™ will be applied on one ovary and fallopian tube.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-45 years at screening.
* Patients undergoing elective laparoscopic surgery involving at least one adnexa.

Exclusion Criteria:

* Pregnant (including ectopic pregnancy) or breastfeeding patient.
* Patients with a documented diagnosis of cancer.
* Patients with a lymphatic, hematologic or coagulation disorder.
* Patients with a known or suspected hypersensitivity to blood, blood products or any constituent of Adhexil™.
* Patients who are immunocompromised, possess autoimmune disorders, or who are routinely taking anticoagulants.
* Patients who have participated in another clinical study within 30 days of enrolment.
* Investigator's opinion that the patient is medically unfit or would be at major risk if enrolled into the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Adhesions will be assessed according to incidence, extent and severity. | 8 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eran Kurman, B.med.Sc, MBA, Study Chair — OMRIX Biopharmaceuticals
Locations (5):
- Richmond, Virginia, United States
- Duisburg, Germany
- Mexico City, Mexico
- Moscow, Russia
- Valencia, Spain